CLINICAL TRIAL: NCT06958549
Title: Management of Multiple Rib Fractures; Role of Nerve Block
Brief Title: Role of Nerve Block in Management of Multiple Rib Fractures
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Kotb, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RIBFRACTURE
Record Dates: First submitted 2025-04-16; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Multiple Rib Fractures
MeSH Terms: interventions — Nerve Block

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nerve block (Active Comparator)
  Interventions: Procedure: Nerve block with Lidocain
- pharmacological analgesics (Active Comparator)
  Interventions: Drug: pharmacological analgesics

INTERVENTIONS:
Procedure: Nerve block with Lidocain — Injection of Lidocaine (7mg/kg) with Epinephrine 1:100000 under Ultrasonographical guidance
  Arms: nerve block
Drug: pharmacological analgesics — Oral Paracetamol (500mg/6hr), IV Ketolac (15mg/6hr) and IV perfelgan (1gm/6hr)
  Arms: pharmacological analgesics

SUMMARY:
* Epidemiology & Impact Thoracic trauma is a common and serious injury worldwide-especially in developing countries-and carries high rates of morbidity and mortality. Complications arise primarily from hypoventilation, which leads to atelectasis, pneumonia, and respiratory failure.
* Key to Reducing Complications: Pain Control Effective analgesia is the cornerstone of preventing respiratory complications. Inadequate pain relief causes patients to splint and hypoventilate, setting the stage for pulmonary collapse and infection.
* Conservative Management
* Analgesics: Systemic pharmacological pain relief remains the mainstay.
* Supportive Measures: Rest, application of ice, and encouragement of deep breathing exercises.
* Incentive Spirometry: Promoted in all patients to maintain lung expansion and ward off atelectasis.
* Regional Anesthesia Techniques

To further improve comfort and respiratory mechanics, ultrasound-guided nerve blocks are employed according to fracture location:

* Serratus Anterior Plane Block for anterolateral rib fractures
* Thoracic Paravertebral Block for posterior rib fractures
* Surgical Intervention Reserved for complex cases-such as flail chest or fractures with risk of organ injury-where stabilization or repair may be necessary.
* Identified Gap Despite these options, thoracic surgeons currently lack a standardized, procedure-specific pain management protocol beyond systemic analgesics, highlighting a need for consensus guidelines that integrate pharmacological and regional techniques.

DETAILED DESCRIPTION:
Thoracic trauma is a major traumatic injury throughout the world, and it has very high incidence in developing countries. Thoracic trauma is often associated with significant morbidity and mortality. Morbidity is due to atelectasis, pneumonia, and respiratory failure as a sequence of hypoventilation.

Most important factor in preventing complications in these patients is pain management. There are different lines of management of multiple rib fractures; conservative therapy is a common line of management which includes appropriate analgesic, rest, and ice.

The use of an incentive spirometer should be encouraged to prevent pulmonary atelectasis and splinting.

Nerve block can also be applied to aid in pain control, surgery may also be a line of management for complicated cases.

The type of nerve block differs according to the site of the fracture; Ultrasound-Guided Serratus Anterior Plane Block is often used for anterolateral rib fractures and Ultrasound-Guided Thoracic Paravertebral Block is used for posterior rib fractures.

The problem here is that ; There is no pain management protocol to be done by thoracic surgeons other than pharmacological analgesics.

This randomized prospective study will be performed in Assiut University Hospitals on two groups of trauma patients, each group is 37 patients; one will undergo nerve block by injection of Lidocaine (7mg/kg) with Epinephrine 1:100000 under ultrasonographical guidance and the other will receive pharmacological analgesics (Oral Paracetamol (500mg/6hr), IV Ketolac (15mg/6hr) and IV perfelgan (1gm/6hr)).

Then improvement in patients pain score, intercostal tube duration in days and total hospital stay in days, patient satisfaction using questionnaire will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* All trauma adult patient (18-70 years) with multiple fracture ribs

Exclusion Criteria:

* Patient with multiple fracture rib with anterior flail segment
* Significant head trauma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Improvement in patients pain score (neumerical score) | day 0, day 1 and day 3

SECONDARY OUTCOMES:
improving intercostal tube duration in days | day 2, day 4 and day 6
improving total hospital stay in days | day 2, day 4 and day 6
improving patient satisfaction (questionnaire) | day 0, day 2, day 4 and day 6

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kring RM, Mackenzie DC, Wilson CN, Rappold JF, Strout TD, Croft PE. Ultrasound-Guided Serratus Anterior Plane Block (SAPB) Improves Pain Control in Patients With Rib Fractures. J Ultrasound Med. 2022 Nov;41(11):2695-2701. doi: 10.1002/jum.15953. Epub 2022 Feb 2. PMID 35106815
- [Background] Yayik AM, Aydin ME, Tekin E, Ulas AB, Ahiskalioglu A. An alternative plane block for multiple rib fractures: Rhomboid Intercostal and Sub-Serratus block (RISS). Am J Emerg Med. 2019 Dec;37(12):2263.e5-2263.e7. doi: 10.1016/j.ajem.2019.158429. Epub 2019 Sep 6. PMID 31526541
- [Background] Hwang EG, Lee Y. Effectiveness of intercostal nerve block for management of pain in rib fracture patients. J Exerc Rehabil. 2014 Aug 31;10(4):241-4. doi: 10.12965/jer.140137. eCollection 2014 Aug. PMID 25210700
- [Background] Easter A. Management of patients with multiple rib fractures. Am J Crit Care. 2001 Sep;10(5):320-7; quiz 328-9. PMID 11548565